CLINICAL TRIAL: NCT05178147
Title: A Feasibility Trial to Evaluate the Use of GraduCheck® in Enabling Experienced Tissue Viability Nurses to Achieve Ideal Sub-Bandage Pressures in Healthy Volunteers
Brief Title: Feasibility Trial of GraduCheck® to Enable Nurses to Achieve Ideal Sub-Bandage Pressures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Whiteley Clinic (Other)
Responsible Party: Principal Investigator, Mark Whiteley, Consultant Venous Surgeon, The Whiteley Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VS-SH-2021-01
Record Dates: First submitted 2021-12-06; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Compression Bandage
Keywords: compression; bandages; wraps; pressure
MeSH Terms: interventions — Compression Bandages

STUDY DESIGN:
Intervention Model Description: To assess the feasibility of using the new GraduCheck® device to enable experienced Tissue Viability Nurses to bandage legs with an optimal pressure profile beneath the bandage, without causing excessive time to be spent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers (Experimental): Volunteers having compression bandages applied to their legs.
  Interventions: Device: Compression bandaging without reference to GraduCheck pressure measurements; Device: Compression bandaging using GraduCheck pressure measurements to monitor compression pressure

INTERVENTIONS:
Device: Compression bandaging without reference to GraduCheck pressure measurements — To apply compression bandages to legs of volunteers without guidance from the Graducheck device (that lies below the bandages) to assess use of the device.
Device: Compression bandaging using GraduCheck pressure measurements to monitor compression pressure — To apply compression bandages to legs of volunteers using the guidance from the Graducheck device (that lies below the bandages) to assess use of the device.

SUMMARY:
The purpose of this study is:

* to evaluate the feasibility of using the GraduCheck® device to optimise the compression profile attained by experienced tissue viability nurses (TVNs) using standard, commonly prescribed, multi-layer bandage systems (Actico, Coban and K2) on healthy volunteers.
* to evaluate the feasibility of using the Graducheck® device to ensure that it does not add excessive time to apply the different sorts of compression bandaging (Actico, Coban and K2) when using the GraduCheck® system to monitor the compression.

DETAILED DESCRIPTION:
This trial is designed to investigate the feasibility of using the GraduCheck® device to achieve optimal compression profiles under compression bandages by experienced TVNs and to check that this does not add excessive time to the bandaging.

This prospective feasibility trial compares the sub-bandage compression profiles achieved by experienced TVNs when applying compression to volunteers without any pressure feedback (hence using experience only), compared with applying compression whilst using the GraduCheck® numerical display for compression feedback during application.

This comparison will be made using three different compression systems on each volunteer. The last system used should be Urgo K2.

The three multi-layer compression bandaging systems will be:

* Actico
* Coban
* Urgo K2

Place of study The study is to be carried out at the Woundcare Consultants Clinic (with a Covid-secure protocol in place).

Healthy Volunteers Twelve (12) healthy volunteers will be recruited.

Assessment of volunteers Before the study commences, any potential volunteer who expresses an interest in joining the study will be given a patient information sheet and a consent form.

Those that have read the patient information sheet and consent form, and still wish to be involved, will be invited in for assessment.

Healthy volunteer participants who fulfil the above criteria (part from those measured at the assessment) will be assessed to by using a Doppler Ability ultrasound device to measure the Ankle Brachial Pressure Index (ABPI), exclude any lower limb ischaemic disease. Healthy volunteer participants must have an ABPI reading between 0.8 and 1.2.

A sphygmomanometer cuff will be placed around the lower legs at the ankle, one after the other, and inflated to 40mmHg. Volunteers will need to be able to tolerate this to be included.

Consent Healthy volunteers who fulfil the inclusion and exclusion criteria (including the assessment of ABPI and cuff inflated around the ankle), to a maximum of 12, will be invited to consent for the study.

The healthy volunteers will have been given an opportunity to discuss any points of the study or consent before signing the consent form.

As part of the consenting process, the healthy volunteers will be informed that they can withdraw at any stage, for any reason, without having to tell the organisers of their reason.

The study protocol The volunteer will be allocated to the TVN who will perform six sequential compression bandage procedures on one of the volunteer's legs, the first three blinded to the GraduCheck® readings and the second three using the GraduCheck®readings to inform the compression being applied. The GraduCheck® compression sensor device will be applied in each of the six sessions.

The time of each compression application will be measured. There will be 12 volunteers treated and 3 TVNs - so each TVN will treat 4 of the volunteers.

The leg to be selected will be on sealed envelope selection (12 sealed envelopes - 6 left and 6 right).

The process will be as follows:

1. - application of first compression system (Actico), blinded to GraduCheck® results:

   * the volunteer is sat in the treatment chair and TVN prepares the Actico compression system and the GraduCheck® compression sensor
   * the GraduCheck® compression system is turned on to record the compression, but positioned so the TVN is unable to see the output
   * when ready, the timer is started
   * the GraduCheck® sensor strip will be applied antero-laterally on the selected limb after the first non-compression (padding) layer is applied. It is important that in volunteers with a significant space from the lateral malleolus to their calf (Achilles tendon) have additional padding placed (at the TVNs discretion).
   * the TVN then applies the Actico compression system as per manufacturer's instructions
   * when the TVN has completed the job the timer is stopped and the time of application is noted
   * the compression profile measured by the GraduCheck® system is recorded by a third party without any communication of the result to the TVN (to prevent any bias before the second two blinded compression system applications)
   * once the figures have been recorded from the GraduCheck® device and the time of the compression application has been noted, the compression system will be removed
   * the healthy volunteer will be asked to stand, stretch and go for a short walk before commencement of the next application
2. - application of second compression system (Coban), blinded to GraduCheck® results:

   * the volunteer is sat in the treatment chair and TVN prepares the Coban compression system and the GraduCheck® compression sensor
   * the GraduCheck® compression system is turned on to record the compression, but positioned so the TVN is unable to see the output
   * when ready, the timer is started
   * the GraduCheck® sensor strip will be applied antero-laterally on the selected limb after the first non-compression (padding) layer is applied. It is important that in volunteers with a significant space from the lateral malleolus to their calf (Achilles tendon) have additional padding placed (at the TVNs discretion).
   * the TVN then applies the Coban compression system as per manufacturer's instructions
   * when the TVN has completed the job the timer is stopped and the time of application is noted
   * the compression profile measured by the GraduCheck® system is recorded by a third party without any communication of the result to the TVN (to prevent any bias before the next blinded compression system application)
   * once the figures have been recorded from the GraduCheck® device and the time of the compression application has been noted, the compression system will be removed
   * the healthy volunteer will be asked to stand, stretch and go for a short walk before commencement of the next application
3. - application of third compression system (Urgo K2), blinded to GraduCheck® results:

   * the volunteer is sat in the treatment chair and TVN prepares the Urgo K2 compression system and the GraduCheck® compression sensor
   * the GraduCheck® compression system is turned on to record the compression, but positioned so the TVN is unable to see the output
   * when ready, the timer is started
   * the GraduCheck® sensor strip will be applied antero-laterally on the selected limb after the first non-compression (padding) layer is applied. It is important that in volunteers with a significant space from the lateral malleolus to their calf (Achilles tendon) have additional padding placed (at the TVNs discretion).
   * the TVN then applies the Urgo K2 compression system as per manufacturer's instructions
   * when the TVN has completed the job the timer is stopped and the time of application is noted
   * the compression profile measured by the GraduCheck® system is recorded by a third party
   * once the figures have been recorded from the GraduCheck® device and the time of the compression application has been noted, the compression system will be removed
   * the healthy volunteer will be asked to stand, stretch and go for a short walk before commencement of the next application
4. - application of first compression system (Actico), using GraduCheck®to inform compression application:

   * the volunteer is sat in the treatment chair and TVN prepares the Actico compression system and the GraduCheck® compression sensor
   * the GraduCheck® compression system is turned on to record the compression, and the output screen turned to the TVN so they can monitor the compression being applied in real time
   * when ready, the timer is started
   * the GraduCheck® sensor strip will be applied antero-laterally on the selected limb after the first non-compression (padding) layer is applied. It is important that in volunteers with a significant space from the lateral malleolus to their calf (Achilles tendon) have additional padding placed (at the TVNs discretion).
   * the TVN then applies the Actico compression system as per manufacturer's instructions, using the output from the GraduCheck® to keep as close as possible to the prescribed pressure of 40 mmHg at the ankle reducing to 20 mmHg just below the knee
   * when the TVN has completed the job the timer is stopped and the time of application is noted
   * the compression profile measured by the GraduCheck® system is recorded
   * once the figures have been recorded from the GraduCheck® device and the time of the compression application has been noted, the compression system will be removed
   * the healthy volunteer will be asked to stand, stretch and go for a short walk before commencement of the next application
5. - application of second compression system (Coban), using GraduCheck® to inform compression application:

   * the volunteer is sat in the treatment chair and TVN prepares the Coban compression system and the GraduCheck® compression sensor
   * the GraduCheck® compression system is turned on to record the compression, and the output screen turned to the TVN so they can monitor the compression being applied in real time
   * when ready, the timer is started
   * the GraduCheck® sensor strip will be applied antero-laterally on the selected limb after the first non-compression (padding) layer is applied. It is important that in volunteers with a significant space from the lateral malleolus to their calf (Achilles tendon) have additional padding placed (at the TVNs discretion).
   * the TVN then applies the Coban compression system as per manufacturer's instructions, using the output from the GraduCheck® to keep as close as possible to the prescribed pressure of 40 mmHg at the ankle reducing to 20 mmHg just below the knee
   * when the TVN has completed the job the timer is stopped and the time of application is noted
   * the compression profile measured by the GraduCheck® system is recorded
   * once the figures have been recorded from the GraduCheck® device and the time of the compression application has been noted, the compression system will be removed
   * the healthy volunteer will be asked to stand, stretch and go for a short walk before commencement of the next application
6. - application of third compression system (Urgo K2), using GraduCheck® to inform compression application:

   * the volunteer is sat in the treatment chair and TVN prepares the Urgo K2 compression system and the GraduCheck® compression sensor
   * the GraduCheck® compression system is turned on to record the compression, and the output screen turned to the TVN so they can monitor the compression being applied in real time
   * when ready, the timer is started
   * the GraduCheck® sensor strip will be applied antero-laterally on the selected limb after the first non-compression (padding) layer is applied. It is important that in volunteers with a significant space from the lateral malleolus to their calf (Achilles tendon) have additional padding placed (at the TVNs discretion).
   * the TVN then applies the Urgo K2 compression system as per manufacturer's instructions, using the output from the GraduCheck® to keep as close as possible to the prescribed pressure of 40 mmHg at the ankle reducing to 20 mmHg just below the knee
   * when the TVN has completed the job the timer is stopped and the time of application is noted
   * the compression profile measured by the GraduCheck® system is recorded
   * if the healthy volunteer is part of the comfort study, then this compression will stay in place and will not be removed
   * if the healthy volunteer is not part of the comfort study, then once the figures have been recorded from the GraduCheck® device and the time of the compression application has been noted, the compression system will be removed
   * the healthy volunteer will be asked to stand, stretch and go for a short walk before being allowed to leave and go home.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Have an ankle brachial pressure index (ABPI) between 0.8-1.2 (at assessment)
* Have no active ulceration

Exclusion Criteria:

* Under the age of 18
* Unable to wear compression bandages of hosiery for any reason
* Unable to walk unaided and at normal speed for at least one mile
* Previous history of deep vein thrombosis
* Have known arterial insufficiency (an ABPI of below 0.8) (at assessment)
* Unable to tolerate a cuff at 40 mmHg around ankle (at assessment)
* Have active ulceration
* Have signs of recent lower limb trauma, active infection, ongoing untreated venous disease, or significant ankle oedema
* Unable to give informed consent
* Pregnant
* Fragile skin that may be damaged whilst trying to apply compression bandaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Pressure profile | 1 day
  Pressure profile obtained under compression bandaging with and without GraduCheck guidance

SECONDARY OUTCOMES:
Time taken to bandage with GraduCheck guidance | 1 day
  Assessment to see how much extra time is used to apply compression with GraduCheck feedback during compression

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Whiteley, MS, Principal Investigator — The Whiteley Clinic Ltd

IPD SHARING:
Plan to Share IPD: No
The results from the study will be presented and submitted of publication in peer-reviewed journals. The results will be presented in table and graphic format. The results from individual volunteers will be included but no personal or identifiable data.

REFERENCES:
- [Background] Bobbink P, Larkin PJ, Probst S. Experiences of Venous Leg Ulcer persons following an individualised nurse-led education: protocol for a qualitative study using a constructivist grounded theory approach. BMJ Open. 2020 Nov 26;10(11):e042605. doi: 10.1136/bmjopen-2020-042605. PMID 33243816
- [Background] Guest JF, Fuller GW, Vowden P. Cohort study evaluating the burden of wounds to the UK's National Health Service in 2017/2018: update from 2012/2013. BMJ Open. 2020 Dec 22;10(12):e045253. doi: 10.1136/bmjopen-2020-045253. PMID 33371051